CLINICAL TRIAL: NCT05017597
Title: Online Cancer-Related Fatigue Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the unversity
Sponsor: Eastern Kentucky University (Other)
Collaborators: University of Dayton (Other)
Responsible Party: Principal Investigator, ANNE FLEISCHER, Professor, Eastern Kentucky University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EasternKU
Record Dates: First submitted 2021-06-10; First posted 2021-08-24 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Neoplasms; Fatigue
Keywords: Function; Fatigue; Occupation; Exercise
MeSH Terms: conditions — Neoplasms; Fatigue; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fatigue management (Experimental): Prescribed exercises by Physical Therapy Problem-Solving Sessions to resume activities that ther person needs to do, wants to do or is expected to do.
  Four online educational modules: What is Cancer-Related Fatigue? Nutrition, Sleep Hygiene and Exercise
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — Exercises completed, and rate of perceived exertion (RPE) will be reviewed during & after each exercise session. Exercises will be modified by either increasing or decreasing the intensity. Decisions will be made based RPE, physical symptoms & any identified barriers or supports. Weeks 1, 3, 5, & 7, Cancer-related fatigue (CRF) education will be assigned. During weeks 2, 4, 6, & 8, CRF education will be reviewed and a plan for how to apply the information will be developed. Participant will be guided through 6 steps of problem solving to address one occupational performance problem identified by participant within Canadian Occupational Performance Measure. Goal & action plan for the week will be shared with the participant electronically. At the beginning of each session, participant will describe progress on previous week action plan. Based on participant's response, either a new goal will be developed or the current one modified..

SUMMARY:
Many individuals who have had cancer experience functional limitations during and after their treatments. The most common side effect from cancer treatment that restricts cancer survivors' completion of daily activities is cancer-related fatigue. Here, we propose to investigate whether an interprofessional approach that targets physiologic, psychologic, and ecological factors will minimize cancer-related fatigue and enhance daily life participation for volunteer cancer survivors living in the community. The interprofessional team will include occupational therapy professor and students from Eastern Kentucky University (EKU), physical therapy and dietitian professors and their students from the University of Dayton, and instructional design instructor from EKU. The approach will include (1) individualized exercise programs-via physical therapy; (2) problem-solving strategies including modifying the environment or activity -via occupational therapy; (3) goal development via physical and occupational therapy; and (4) cancer-related fatigue education via instructional design. We hypothesize that this approach will result in participants experiencing less fatigue, increasing their mobility, improving their quality of life, and being more satisfied with how they perform daily activities.

DETAILED DESCRIPTION:
Setting: Virtual environment

1. Evaluation and weekly meetings will be provided through Zoom® conferencing system provided by EKU or University of Dayton.
2. Educational and Exercise Videos will be accessed within an individual webpage for each participant within the study's website.

Research Design Pre-test/Post-test quasi-experimental design without a control group. This research design will allow us to assess if there is a change in the level of fatigue, mobility, quality of life, and/or perceived performance and satisfaction of important activities Screening Individuals who are interested in participating will contact the Occupational Therapy professor--principal investigator (PI) or Physical Therapy professor-collaborator (CL). PI or CL will contact the potential participant either by telephone or email. Within this initial communication, the potential participant will be provided with the following information: time commitment, type of evaluations, and intervention. If the participant continues to be interested, an electronic inclusion criteria screen will be sent. If all inclusion criteria are met, PI or CL will ask the participant for their physician contact information so a medical release form can be sent to them.

Physician medical release A release form will be faxed, sent electronically, or mailed to participant's oncology or primary care provider. Once this signed release is received, we will send an electronic version of the informed consent to the potential participant and schedule a time to review it and a tentative time for the initial evaluation.

Initial, Weekly, 4-week, and 8-week Standard of Care Cancer Survivor Evaluations Initial Evaluations After the participant agrees to take part in the study and signs the informed consent, the initial evaluation including questionnaires and physical therapy and occupational therapy assessments within one to two visits will be administered by physical therapy and occupational therapy students (PTSI and OTSI). Assessments will be recorded and reviewed by the supervising therapy professor to ensure assessments are performed using standardized methods. After the assessment eight weekly meetings will be schedule.

* Estimated length of weekly meeting is 20-30 minutes.
* Each exercise session is 30-45 minutes in length depending on which level of exercise the participant is completing. The participant will complete 3 sessions each week.
* Each participant will be provided their own webpage, which can only be accessed by them and the researchers. Within the webpage, the researchers will store the prescribed exercise program, including handouts, video and exercise log, and the problem-solving session goals and action plans. Links to the Cancer-Related Fatigue (CRF) educational modules, as they are assigned to the participant will be posted as well.

ELIGIBILITY:
Inclusion Criteria:

* Completed treatment for a cancer diagnosis within 5 years of enrollment
* Access to mobile device or computer
* Basic computer or mobile device skills
* Experience a significant level of fatigue defined as >= 4 on 0-10 scale using the One-item Fatigue Scale.

Exclusion Criteria:

* Currently undergoing chemotherapy or radiation treatment
* Unwilling to participate in an exercise program
* Have metastatic cancer (Stage 4)
* Do not have physician consent to participate in the exercise program
* Unable to follow verbal or written assessment instructions
* Non-English speaking.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in Fatiue Level: Brief Fatigue Inventory | Change from Baseline measure at 4 weeks
  This 9-item scale assesses the severity and interference of fatigue on a 0 (no fatigue) to 10 (greatest fatigue) scale
Change in Fatiue Level: Brief Fatigue Inventory | Change from 4 week measure at 8 weeks
  This 9-item scale assesses the severity and interference of fatigue on a 0 (no fatigue) to 10 (greatest fatigue) scale
Perceived Functional Change: Canadian Occupational Performance Measure | Change from Baseline measure at 4 weeks
  a semi-structured interview to understand the routine activities that the participant completes daily, specifically their self-care, leisure, and social activities. The participant rates the importance of each of the activities using a 0 to 10 scale. Zero indicates "no importance" and 10 indicates "very important." Then the participant rates their perception of how well they currently perform each of the important activities and how satisfied they are with their performance using a 0 to 10 scale. Zero indicates that "they are not able to perform" or "they are not satisfied" and 10 indicates that "they are able to perform the activity well" or "they are very satisfied." This is repeated for how satisficed with how they currently perform each important activity.
Perceived Functional Change: Canadian Occupational Performance Measure | Change from 4 week measure at 8 weeks
  a semi-structured interview to understand the routine activities that the participant completes daily, specifically their self-care, leisure, and social activities. The participant rates the importance of each of the activities using a 0 to 10 scale. Zero indicates "no importance" and 10 indicates "very important." Then the participant rates their perception of how well they currently perform each of the important activities and how satisfied they are with their performance using a 0 to 10 scale. Zero indicates that "they are not able to perform" or "they are not satisfied" and 10 indicates that "they are able to perform the activity well" or "they are very satisfied." This is repeated for how satisficed with how they currently perform each important activity.

SECONDARY OUTCOMES:
One Item Fatigue Scale | Change from baseline measure at 8 weeks
  Participants answer the following question: "How would you rate your fatigue on a scale of 0 to10 with 0 being 'no fatigue' and 10 being the 'worst possible fatigue'
FACIT-Fatigue | Change from Baseline measure at 8 weeks
  This 40-item 5-point Likert scale evaluates quality of life in individuals with fatigue as measured in 5 domains: physical, social/family, emotional, functional well-being, and fatigue. Higher scores reflect greater quality of life
6-minute walk test | Change from baseline measure at 4 weeks
  Participants will complete a 6-minute walk at their chosen pace, using assistive devices if needed and with permitted standing rest breaks. Participants will be required to measure the length of a hallway, sidewalk, or driveway where they will be walking. They will then walk for 6 minutes. Participants will report the distance walked as well as the number of rest breaks taken during the 6 minutes.
6-minute walk test | Change from 4 week measure at 8 weeks
  Participants will complete a 6-minute walk at their chosen pace, using assistive devices if needed and with permitted standing rest breaks. Participants will be required to measure the length of a hallway, sidewalk, or driveway where they will be walking. They will then walk for 6 minutes. Participants will report the distance walked as well as the number of rest breaks taken during the 6 minutes.
30-second Sit to Stand | Change from baseline measure at 4 weeks
  Participants are seated in a standard height fixed chair without armrests, which is placed against a wall. They will move from sitting to standing and back to sitting position, with arms crossed against chest. The number of complete stands and sits (1 repetition) will be counted by the investigator and the participant within 30 seconds
30-second Sit to Stand | Change from 4 week measure at 8 weeks
  Participants are seated in a standard height fixed chair without armrests, which is placed against a wall. They will move from sitting to standing and back to sitting position, with arms crossed against chest. The number of complete stands and sits (1 repetition) will be counted by the investigator and the participant within 30 seconds
Borg Perceived Exertion 6-20 scale | Change from baseline measure to 4 weeks
  This scale allows participants to rate their perceived exertion during physical activity. Patients will be instructed to rate their level of exertion during their home exercise program and at the conclusion of each session. This will be recorded on their weekly exercise log.
Borg Perceived Exertion 6-20 scale | Change from 4 week measure to 8 weeks
  This scale allows participants to rate their perceived exertion during physical activity. Patients will be instructed to rate their level of exertion during their home exercise program and at the conclusion of each session. This will be recorded on their weekly exercise log.

OTHER OUTCOMES:
Maximum heart rate and target heart rate range | Baseline
  The investigator will calculate the participant's maximum heart rate using the formula 207-.70(age)= maximum heart rate. The prescribed exercise intensity will be based on this calculation. The investigator will then instruct the participant on how to measure their heart rate to monitor their exercise intensity during exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fleischer, Ph.D, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Only researchers involved in this study, who have been approved by the Institutional Review Board, will have access to the data.

REFERENCES:
- [Background] Bronfenbrenner U. Toward an experimental ecology of human development. American Psychologist. 1977. 32: 513-531
- [Background] Champion VL, Wagner LI, Monahan PO, Daggy J, Smith L, Cohee A, Ziner KW, Haase JE, Miller KD, Pradhan K, Unverzagt FW, Cella D, Ansari B, Sledge GW Jr. Comparison of younger and older breast cancer survivors and age-matched controls on specific and overall quality of life domains. Cancer. 2014 Aug 1;120(15):2237-46. doi: 10.1002/cncr.28737. Epub 2014 May 28. PMID 24891116
- [Background] Du S, Hu L, Dong J, Xu G, Jin S, Zhang H, Yin H. Patient education programs for cancer-related fatigue: A systematic review. Patient Educ Couns. 2015 Nov;98(11):1308-19. doi: 10.1016/j.pec.2015.05.003. Epub 2015 May 23. PMID 26072422
- [Background] Gellish RL, Goslin BR, Olson RE, McDonald A, Russi GD, Moudgil VK. Longitudinal modeling of the relationship between age and maximal heart rate. Med Sci Sports Exerc. 2007 May;39(5):822-9. doi: 10.1097/mss.0b013e31803349c6. PMID 17468581
- [Background] Hegel MT, Lyons KD, Hull JG, Kaufman P, Urquhart L, Li Z, Ahles TA. Feasibility study of a randomized controlled trial of a telephone-delivered problem-solving-occupational therapy intervention to reduce participation restrictions in rural breast cancer survivors undergoing chemotherapy. Psychooncology. 2011 Oct;20(10):1092-101. doi: 10.1002/pon.1830. Epub 2010 Sep 5. PMID 20821373
- [Background] Hong Y, Pena-Purcell NC, Ory MG. Outcomes of online support and resources for cancer survivors: a systematic literature review. Patient Educ Couns. 2012 Mar;86(3):288-96. doi: 10.1016/j.pec.2011.06.014. Epub 2011 Jul 27. PMID 21798685
- [Background] Hoybye MT, Dalton SO, Deltour I, Bidstrup PE, Frederiksen K, Johansen C. Effect of Internet peer-support groups on psychosocial adjustment to cancer: a randomised study. Br J Cancer. 2010 Apr 27;102(9):1348-54. doi: 10.1038/sj.bjc.6605646. PMID 20424614
- [Background] Lindahl-Jacobsen L, Hansen DG, Waehrens EE, la Cour K, Sondergaard J. Performance of activities of daily living among hospitalized cancer patients. Scand J Occup Ther. 2015 Mar;22(2):137-46. doi: 10.3109/11038128.2014.985253. Epub 2015 Jan 12. PMID 25580840
- [Background] Lyons KD, Newman RM, Kaufman PA, Bruce ML, Stearns DM, Lansigan F, Chamberlin M, Bartels SJ, Whipple J, Hegel MT. Goal Attainment and Goal Adjustment of Older Adults During Person-Directed Cancer Rehabilitation. Am J Occup Ther. 2018 Mar/Apr;72(2):7202205110p1-7202205110p8. doi: 10.5014/ajot.2018.023648. PMID 29426388
- [Background] Ma Y, He B, Jiang M, Yang Y, Wang C, Huang C, Han L. Prevalence and risk factors of cancer-related fatigue: A systematic review and meta-analysis. Int J Nurs Stud. 2020 Nov;111:103707. doi: 10.1016/j.ijnurstu.2020.103707. Epub 2020 Jul 11. PMID 32920423
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Silver JK, Baima J, Newman R, Galantino ML, Shockney LD. Cancer rehabilitation may improve function in survivors and decrease the economic burden of cancer to individuals and society. Work. 2013;46(4):455-72. doi: 10.3233/WOR-131755. PMID 24125901
- [Background] Owen JE, Klapow JC, Roth DL, Shuster JL Jr, Bellis J, Meredith R, Tucker DC. Randomized pilot of a self-guided internet coping group for women with early-stage breast cancer. Ann Behav Med. 2005 Aug;30(1):54-64. doi: 10.1207/s15324796abm3001_7. PMID 16097906
- [Background] Salzer MS, Palmer SC, Kaplan K, Brusilovskiy E, Ten Have T, Hampshire M, Metz J, Coyne JC. A randomized, controlled study of Internet peer-to-peer interactions among women newly diagnosed with breast cancer. Psychooncology. 2010 Apr;19(4):441-6. doi: 10.1002/pon.1586. PMID 19484712
- [Background] Smith TM, Broomhall CN, Crecelius AR. Physical and Psychological Effects of a 12-Session Cancer Rehabilitation Exercise Program. Clin J Oncol Nurs. 2016 Dec 1;20(6):653-659. doi: 10.1188/16.CJON.653-659. PMID 27857248
- [Background] Yun YH, Lee KS, Kim YW, Park SY, Lee ES, Noh DY, Kim S, Oh JH, Jung SY, Chung KW, Lee YJ, Jeong SY, Park KJ, Shim YM, Zo JI, Park JW, Kim YA, Shon EJ, Park S. Web-based tailored education program for disease-free cancer survivors with cancer-related fatigue: a randomized controlled trial. J Clin Oncol. 2012 Apr 20;30(12):1296-303. doi: 10.1200/JCO.2011.37.2979. Epub 2012 Mar 12. PMID 22412149
- [Background] Zabit F, Iyigun G. A comparison of physical characteristics, functions and quality of life between breast cancer survivor women who had a mastectomy and healthy women. J Back Musculoskelet Rehabil. 2019;32(6):937-945. doi: 10.3233/BMR-181362. PMID 31282398